CLINICAL TRIAL: NCT05889338
Title: Impact of Adalimumab Therapy on Quality of Life of Patients With Severe Psoriasis
Brief Title: Effect of Adalimumab Therapy on Psoriasis Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shimaa Fawzy Abdelhalim, Dermatology resident at Gehina Hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-04-26MS_
Record Dates: First submitted 2023-05-11; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Psoriasi
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case: adults with severe psoriasis treated by adalimumab therapy. (Active Comparator)
  Interventions: Drug: adalimumab and methotrexate
- Control: adults with severe psoriasis treated by methotrexate therapy. (Active Comparator)
  Interventions: Drug: adalimumab and methotrexate

INTERVENTIONS:
Drug: adalimumab and methotrexate — Adult patients (> 18 years) with severe psoriasis who will start treatment with either adalimumab or methotrexate

SUMMARY:
to evaluate the impact of adalimumab therapy on quality of life in patient with severe psoriasis.

DETAILED DESCRIPTION:
to evaluate the impact of adalimumab therapy against methotrexate therapy on quality of life in patient with severe psoriasis and follow up after 24 week by A- Medical history age, sex, marital state, occupation, educational level and family history. dermatologic history: onset, course, duration. B- Complete dermatologic examination

C- Psoriasis Area and Severity Index (PASI) score:

The scoring involves rating the symptoms of psoriasis from none to very severe and estimating the percentage of the body that they affect.The range of absolute PASI scores is 0-72, with higher scores indicating a greater severity of psoriasis. A score of 0 indicates no psoriasis, while a score higher than 10 suggests severe psoriasis. The scoring system includes a section for intensity and another for body coverage .The score will be evaluated before treatment, at week 12 and at week 24.

D- Dermatology Life Quality Index (DLQI):

It is self-reported questionnaire . It has been translated to >110 languages. Measurement properties of the DLQI, such as validity, reliability, and responsiveness to change were reported. It is widely used in both clinical practice and research settings, including randomized controlled trials, patient registries, and national treatment and reimbursement guidelines . The study will depend on the Arabic Tunisian version of the DLQI questionnaire . DLQI consists of 10 questions related to symptoms, feelings, daily activities, leisure, work, personal relationships and the effects of treatment on daily life within the past week. Scores can range from 0 to 30, with higher scores representing worse quality of life . The questionnaire will be answered by all participant before initiation of treatment, at week 12 and at week 24 of treatment.

ELIGIBILITY:
Inclusion Criteria:

.Adult patients (> 18 years) with severe psoriasis who will start treatment with either adalimumab or methotrexate.

Exclusion Criteria:

.Pregnancy or lactation. .Chronic liver or renal disease. .History of tuberculosis. .Cancer and blood disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index | 6 month
  The scoring involves rating the symptoms of psoriasis from none to very severe and estimating the percentage of the body that they affect.The range of absolute PASI scores is 0-72, with higher scores indicating a greater severity of psoriasis. A score of 0 indicates no psoriasis, while a score higher than 10 suggests severe psoriasis. The scoring system includes a section for intensity and another for body coverage .

SECONDARY OUTCOMES:
Dermatology Life Quality Index | 6 month
  It is self-reported questionnaire . It has been translated to >110 languages. Measurement properties of the DLQI, such as validity, reliability, and responsiveness to change were reported. It is widely used in both clinical practice and research settings, including randomized controlled trials, patient registries, and national treatment and reimbursement guidelines . The study will depend on the Arabic Tunisian version of the DLQI questionnaire . DLQI consists of 10 questions related to symptoms, feelings, daily activities, leisure, work, personal relationships and the effects of treatment on daily life within the past week. Scores can range from 0 to 30, with higher scores representing worse quality of life .

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rencz F, Szabo A, Brodszky V. Questionnaire Modifications and Alternative Scoring Methods of the Dermatology Life Quality Index: A Systematic Review. Value Health. 2021 Aug;24(8):1158-1171. doi: 10.1016/j.jval.2021.02.006. Epub 2021 Apr 21. PMID 34372982
- [Background] Frenzel A, Schirrmann T, Hust M. Phage display-derived human antibodies in clinical development and therapy. MAbs. 2016 Oct;8(7):1177-1194. doi: 10.1080/19420862.2016.1212149. Epub 2016 Jul 14. PMID 27416017
- [Background] van der Kraaij G, Busard C, van den Reek J, Menting S, Musters A, Hutten B, de Rie M, Ouwerkerk W, van Bezooijen SJ, Prens E, Rispens T, de Vries A, de Jong E, de Kort W, Lambert J, van Doorn M, Spuls P. Adalimumab with Methotrexate vs. Adalimumab Monotherapy in Psoriasis: First-Year Results of a Single-Blind Randomized Controlled Trial. J Invest Dermatol. 2022 Sep;142(9):2375-2383.e6. doi: 10.1016/j.jid.2022.01.033. Epub 2022 Mar 8. PMID 35276223
- [Background] Matsui T, Umetsu R, Kato Y, Hane Y, Sasaoka S, Motooka Y, Hatahira H, Abe J, Fukuda A, Naganuma M, Kinosada Y, Nakamura M. Age-related trends in injection site reaction incidence induced by the tumor necrosis factor-alpha (TNF-alpha) inhibitors etanercept and adalimumab: the Food and Drug Administration adverse event reporting system, 2004-2015. Int J Med Sci. 2017 Jan 15;14(2):102-109. doi: 10.7150/ijms.17025. eCollection 2017. PMID 28260984